CLINICAL TRIAL: NCT03194295
Title: Activating Personal Network Support in Treatment Seeking Substance Users
Brief Title: Activating Community Support for Substance Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00130614; 1R34DA042320-01A1 (NIH)
Record Dates: First submitted 2017-02-24; First posted 2017-06-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Substance Use Disorders
Keywords: Drug-free community support; Methadone maintenance; Social networks
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Meets criteria of a phase II non-pharmacological treatment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Support Intervention (Experimental): Participants randomized to this condition will be scheduled to attend a 12-week (1x/wk for one hour) manual-guided Community Support Intervention Group, which requires methadone maintenance treatment (MMT) participants to attend the group with a drug-free family member or friend (community support person; CSP).
  Interventions: Behavioral: Community Support Intervention Group
- Standard Care (Active Comparator): Participants randomized to this condition will be scheduled to attend a 12-week (1x/wk for one hour) manual-guided Substance Use Disorder Educational Group as an attention-control for the intervention described in the experimental condition.
  Interventions: Behavioral: Substance Use Disorder Educational Group

INTERVENTIONS:
Behavioral: Community Support Intervention Group — This 12-week community support intervention is designed to activate and harness the powerful influences of drug-free family and friends to enhance recovery support and participation in community activities. Addiction Treatment Services (ATS) participants and their CSPs will be directed to participate in recovery-oriented community activities together 2 times per week and work together toward developing regular drug-free social support for the ATS participant. The group provides an opportunity for both the participant and CSP to discuss their experiences participating in the scheduled activities. For those electing not to engage in community activities, problem-solving strategies will be used to remove obstacles to participation, with other group members providing support and encouragement.
  Arms: Community Support Intervention
Behavioral: Substance Use Disorder Educational Group — This 12-week educational group is designed as an attention-control group. Group topics include: 1) definition of substance dependence, 2) the disease model, 3) medical aspects, 4) mood, 5) personality, 6) self-esteem, 7) relapse prevention, 8) HIV/AIDS, 9) anger, 10) negative thinking, 11) nutrition, and 12) assertiveness. Participants will be assigned 2 homework assignments each week based on the topic.
  Arms: Standard Care

SUMMARY:
Efforts to improve methadone maintenance outcomes are often thwarted by strong social networks that reinforce substance use and other risk behaviors. The proposed study the feasibility and preliminary efficacy of a practical community support intervention that employs an alteration model of social network change. The intervention works with patients and at least one drug-free family or friend to support participation in community activities designed to mobilize recovery support and expand personal drug-free social networks.

DETAILED DESCRIPTION:
Opioid-dependent individuals in methadone maintenance have high rates of illicit drug and alcohol use. The individual and public health concerns of poorly and partially treated substance use include social, medical, psychiatric, and healthcare costs. Efforts to improve outcomes are often thwarted by strong social networks that reinforce substance use and other high-risk drug use and sexual behaviors. Many urban substance users lack the financial resources to simply move away from adverse community influences. While clinical providers are well aware of the power of social network influences, existing research provides relatively little direction about how to help substance users change "people, places, and things." An under-explored strategy to achieve this desired outcome is to mobilize social support found in the personal social networks of people with substance use disorder. A considerable amount of research demonstrates that people with substance use disorder routinely have drug-free family or friends in their social networks, and that these individuals are terribly underutilized for supporting recovery efforts. Social support is reliably associated with good health behaviors and more positive and sustained substance abuse treatment outcomes. The inclusion of drug-free family and friends also provides a pathway to modify social networks by facilitating activity with other drug-free people within and outside of the patient's social network. This type of work supports an alteration model of network change. This protocol uses an alteration model to develop a promising 12-week community support intervention designed to activate and harness the powerful influences of drug-free family and friends to enhance recovery support and participation in community activities. This highly structured and manual-guided therapeutic group works with patients and at least one drug-free family member or friend (community support person -- CSP) to expand the quantity and quality of the patients' drug-free social network, and to reduce and eliminate interactions with active drug users. This outcome is achieved via a series of "homework" assignments that require the patient and CSP to participate together in two drug-free activities per week that include the presence of other drug-free individuals (e.g., Narcotics Anonymous (NA)/Alcoholics Anonymous (AA), religious activities), and to discuss their experiences within the group setting. This intervention will be compared to Standard Care that includes a substance abuse education group with weekly homework. Specific aims evaluate feasibility outcomes and the extent to which the intervention supports an alteration model. Short-term efficacy will be assessed using measures of perceived social support and network support for abstinence. Secondary outcomes will evaluate substance use and psychosocial outcomes. Data will support a larger-scale randomized clinical trial (RCT) better isolating the clinical benefits of activating existing social support and facilitating community involvement.

ELIGIBILITY:
Inclusion Criteria (for the ATS participant):

* ATS treatment participation of more than 4-weeks
* Submission of at least one drug-positive urine sample
* Expressed willingness to include a drug-free support person in treatment

Exclusion Criteria (for the ATS participant):

* Pregnancy
* Acute medical problem that requires immediate and intense medical management (e.g., AIDS defining illness; unstable diabetes)
* Presence of a formal thought disorder, delusions, hallucinations, or imminent risk of harm to self or others
* Unable to read.

Exclusion Criteria (for the CSPs)

* Submission of a drug-positive urine sample
* Pregnancy
* Acute medical problem that requires immediate and intense medical management (e.g., AIDS defining illness; unstable diabetes)
* Presence of a formal thought disorder, delusions, hallucinations, or imminent risk of harm to self or others
* Unable to read.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Perceived social support for designated CSP as assessed by the Quality of Relationships Inventory (QRI) "support scale" | Monthly for 3 months
  The investigators anticipate that Community Support (vs. Standard Care) participants will enjoy greater levels of perceived social support (QRI "support" scale, a continuous measure) at the 3-month evaluation. Mixed model analyses will be used to evaluate condition differences over time (Baseline, Months 1-3). The two remaining QRI subscales ("conflict"; "depth") will also be examined using a similar analytic approach.
Behavioral and attitudinal support for abstinence as assessed by the IPA | Monthly for 3 months
  The investigators anticipate Community Support (vs. Standard Care) participants will enjoy more Behavioral and Attitudinal support for Abstinence (IPA scales; continuous measures) over the 3-month evaluation. Mixed model analyses will be used to evaluate condition differences over time (Baseline, Month 3). The remaining IPA subscales (Social Support for Drug Use; Behavioral Support for Drug Use; Attitudinal Support for DrugUse) will be examined in secondary analyses using a similar approach.

SECONDARY OUTCOMES:
Substance use and problem severity as assessed by urinalysis testing and Addiction Treatment Index (ASI) composite scores | Monthly for 3 months
  The investigators anticipate Community Support (vs. Standard Care) participants will have lower rates of "any" drug-positive urine samples (i.e., opioid, cocaine, sedatives, and/or cannabis) over the 3-month evaluation.
  Drug-positive urine samples will be treated as a dichotomous variable. Generalized estimating equation (GEE) analysis will be used to evaluate condition differences over time (Baseline, Months 1-3). Specific classes of drugs (opioid, cocaine, sedative, cannabis positive urinalysis tests) will be examined using a similar analytic approach. Secondary analyses will use mixed model analyses to evaluate condition differences in ASI self-report drug composite scores over time (Baseline, Months 1-3). The remaining ASI composite scores will be examined using a similar approach.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kidorf, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kidorf M, Peirce J, Brooner RK, Yan H, Latkin C. Feasibility and preliminary efficacy of a community support intervention for people with opioid use disorder. Am J Addict. 2023 Nov;32(6):554-562. doi: 10.1111/ajad.13457. Epub 2023 Aug 8. PMID 37553840